CLINICAL TRIAL: NCT06990659
Title: CHOC - Implémentation et évaluation d'un Parcours de Soin Ambulatoire Pour Les Patients traités Par Voie Intra-artérielle d'un Cancer Primitif du Foie : Essai Multicentrique contrôlé randomisé
Brief Title: Outpatient Care Pathway for Patients Treated Intra-arterially for Primary Liver Cancer
Acronym: CHOC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Université Paris Cité (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 49RC23_0306; 2024-A02727-40 (Other: ANSM)
Record Dates: First submitted 2025-04-24; First posted 2025-05-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hepato Cellular Carcinoma (HCC)
Keywords: ambulatory care; hospitalization; Hepato cellular carcinoma; Patient satisfaction; randomized trial; chemoembolization; radioembolization
MeSH Terms: conditions — Patient Satisfaction | interventions — Ambulatory Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Ambulatory care (Experimental): Ambulatory care : Outpatient management of radiological treatment for HCC
  Interventions: Other: Ambulatory care
- Arm Conventional inpatient care (Other): Conventional inpatient care : Conventional inpatient management for radiological treatment of HCC
  Interventions: Other: Conventional inpatient care

INTERVENTIONS:
Other: Ambulatory care — Patients with Hepato cellular carcinoma (HCC) treated by chemo-embolization (CEH) or radioembolization (REH) are managed on an outpatient basis: hospitalization in an outpatient unit, followed by systematic telephone and on-demand nursing follow-up for 48 hours for REH and 72 hours for CEH. A dedicated re-hospitalization circuit has also been set up in the event of complications.
  Arms: Arm Ambulatory care
Other: Conventional inpatient care — Patients with Hepato cellular carcinoma (HCC) treated by chemo-embolization (CEH) or radioembolization (REH) are managed on an inpatient basis: conventional hospitalization.
  Arms: Arm Conventional inpatient care

SUMMARY:
Randomized trial comparing two care organizations (outpatient versus conventional inpatient care) using a mixed method (quantitative and qualitative data and analysis).

The protocol involves randomization between an ambulatory group and a conventional hospitalization group. Patients will be monitored for 7 months to assess satisfaction, complications and treatment efficacy. A qualitative study will be carried out to understand the obstacles and facilitate implementation of the ambulatory pathway. A medico-economic analysis will accompany this study to assess the financial impact of adopting the ambulatory pathway. The expected results will help determine the best management strategy for these patients.

The study's hypotheses are that performing intra-arterial treatments for primary liver cancer on an outpatient basis, combined with telephone follow-up, will improve patient satisfaction with their care, and that analysis of the implementation of this outpatient pathway will help improve the pathway and facilitate its implementation at other sites, by identifying obstacles and solutions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* HCC or CCi diagnosed according to the criteria of the European Association for the Study of the Liver (2024) or histologically proven.
* HCC or CCi naive to intra-arterial treatment. HCC may have been previously treated with other non-intra-arterial therapies. Other HCC may have been previously treated but not with intra-arterial therapy.
* If HCC treatment is proposed at a Multidisciplinary Consultation Meeting (RCP):
* Patient Child-Pugh < B8
* Single or multiple HCC
* Absence of lobar or truncal portal obstruction
* Absence of bile duct dilatation
* If treatment by REH proposed in RCP:
* Absence of truncal portal tumor invasion
* Uni-lobar tumor invasion (except for centrohepatic CCi)
* Total bilirubin < 20 mg/l (or 35 µmol/L)
* Patient affiliated to or benefiting from a social security scheme
* Patient having signed an informed consent form

Exclusion Criteria:

* Technical contraindication or morphological elements of predictable technical difficulty
* Chronic renal insufficiency (Clairance < 30 ml/min)
* Known allergy to a contrast agent or chemotherapy agent
* Patient unable to be a candidate for outpatient management
* Patient previously included in the study
* Patient who, for psychological, social, family or geographical reasons, could not be regularly monitored, patient who, for psychological, social, family or geographical reasons, could not be followed regularly
* Concomitant disease or severe uncontrolled clinical situation
* Severe uncontrolled infection
* Pregnant, breast-feeding or parturient woman
* Person deprived of liberty by judicial or administrative decision
* Person under compulsory psychiatric care
* Person under a legal protection measure
* Person unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall patient satisfaction | 72 hours after treatment procedure
  EORTC PATSAT-C33 questionnaire. All items are scored 1 (bad) to 5 (excellent). The total score measures range in score from 0 to 100. A high score represents a high level of satisfaction with care / perceived care quality.

SECONDARY OUTCOMES:
Acceptability (quantitative) | At inclusion visit (pre-treatment)
  Proportion of consenting patients and description of refusals
Acceptability (qualitative) | At inclusion visit (pre-treatment)
  Thematic analysis of individual research interviews with a sample of patients included in both arms of the study.
4. Adoption (quantitative) | 32 months
  Number of outpatient courses completed compared with the number of scheduled courses; number of candidate, open and active centers.
Adoption (qualitative) | 36 months
  Thematic analysis of verbatims collected during focus groups with centers
Relevance (reasons for refusal) | 24 months
  Characteristics of patients whose inclusion in the protocol was refused by the patient/carer.
Relevance (patient expectations) | 36 months
  Thematic content analysis of verbatims collected during individual research interviews with patients in both arms, in order to understand the patient experience throughout the treatment period, and to identify needs and expectations in terms of post-intervention follow-up in both groups.
Feasibility of outpatient care | One year after the end of inclusions
  Proportion of outpatient treatments planned and then cancelled, reasons for non-implementation, perception of obstacles and facilitators via individual interviews and focus groups with caregivers.
Scope (Quantitative) | One year after the end of inclusions
  Patient-related factors associated with ambulatory care pathway failure (Indication; Techniques; Tolerance of organization).
Scope (Qualitative for centers) | One year after the end of inclusions
  thematic analysis of verbatims collected in the focus group, focusing on elements identified by caregivers as having contributed to organizational changes to enable implementation of the ambulatory pathway. Elements perceived as obstacles to change will also be identified and analyzed by theme
Scope (Qualitative for patients) | One year after the end of inclusions
  thematic analysis of verbatims collected during post-treatment interviews, focusing on elements identified by patients as having contributed to their continued health after returning home. Elements relating to improvements to be made to the ambulatory care pathway will also be recorded and analyzed by theme
Comparing the organizations (Comfort and satisfaction) | day of surgery, evening after surgery and 10 days after treatment
  Visual analogue scale (VAS) for pain : 0 ('no pain') to 10 ('pain as bad as it could possibly be')
Comparing the organizations (Comfort and satisfaction) | 72 hours after treatment
  Quality Of Life Questionnaire - Satisfaction with Cancer Care - Core questionnaire (EORTC QLQ-PATSAT-C33) for all and specific complementary outpatient module (OUT-PATSAT7) for the outpatient group.
  Items are rated from 1 (bad) to 5 (Excellent)
Comparing the organizations (Quality of life) | At inclusion visit (pre-treatment), Day 7, Month2/Month3 visit
  Medical Outcome Study Short Form 12 (SF-12) A score >50 indicates above-average health-related quality of life
Comparing the organizations (General condition) | At inclusion visit (pre-treatment), Month2/Month3 visit
  Patient's general condition assessed by clinical status (Eastern Cooperative Oncology Group ECOG) from 0 (Fully active, able to carry on all pre-disease performance without restriction) to 5 (dead)
Comparing the organizations (Complications) | Month 6
  Complications according to the Common Terminology Criteria for Adverse Events (CTCAE) V5.0.5 Items from 1 (mild) to 5 (death)
Comparing the organizations (Technical succes) | Month2/Month3 visit, Month 6
  Technical success defined by completion of the planned procedure. Tumor response according to Response Evaluation Criteria in Solid Tumors (mRECIST) and Liver Imaging Reporting and Data System (LIRADS)
Factors for patient satisfaction (HADS) | Inclusion, Admission before surgery and 72 hours after treatment
  Anxiety and depression scale (HADS)
Factors for patient satisfaction (Disease characteristics) | At inclusion visit (pre-treatment)
  Barcelona Clinic Liver Cancer (BCLC) classification stage, sarcopenia (based on imaging).
Factors for patient satisfaction (Treatment characteristics) | Day of treatment procedure
  1. for hepatic chemoembolization (CEH): selectivity, number of segments treated, % of chemotherapy injected, additional embolization;
  2. for radioembolization (REH): number of injection sites;
  3. for all: procedure duration, center volume, operator volume, treatment line, combination treatment.
Factors for patient satisfaction (socioeconomic) | At inclusion visit (pre-treatment)
  Socioeconomic level
Factors for patient satisfaction (travel) | At inclusion visit (pre-treatment)
  Home-hospital travel time
Factors for patient satisfaction (comorbidities) | At inclusion visit (pre-treatment)
  Comorbidities
Factors for patient satisfaction (ECOG) | At inclusion visit (pre-treatment)
  Clinical status (ECOG)
Factors for patient satisfaction (Quality of life) | At inclusion visit (pre-treatment), Day 7, Month 2/Month3
  Questionnary of quality of life = Medical Outcome Study Short Form 12 (SF-12)
Total cost of each treatment pathway | From day of treatment to Month 2/Month 3 visit
  From the community, health insurance and hospital perspective (depending on the type of treatment received)
Budgetary impact | 5 years after study
  Annual and cumulative 5-year budgetary impact of changing clinical practices towards outpatient management of patients treated intra-arterially for hepatocellular carcinoma, from a health insurance perspective

CONTACTS AND LOCATIONS:
Overall Officials: Christophe AUBE, Pr, Principal Investigator — University Hospital, Angers
Locations (16):
- France (16):
  - University hospital of Amiens, Amiens
  - University hospital of Angers, Angers
  - University hospital of Besançon, Besançon
  - Hospital of Avicennes (AP-HP), Bobigny
  - University hospital of Brest, Brest
  - University hospital of Clermont-Ferrand, Clermont-Ferrand
  - Hospital of Beaujon (AP-HP), Clichy
  - Hospital of Vendée, La Roche-sur-Yon
  - University hospital of Grenoble-Alpes, La Tronche
  - University hospital of Montpellier, Montpellier
  - Nantes, Nantes
  - University hospital of Nice, Nice
  - Hospital of Pitié-Salpétrière (AP-HP), Paris
  - Hospital of Cochin (AP-HP), Paris
  - Univesity hospital of Bordeaux, Pessac
  - Institut Gustave Roussy (IGR), Villejuif

IPD SHARING:
Plan to Share IPD: No